CLINICAL TRIAL: NCT04155086
Title: "Fetal Aneuploidy Screening (21, 18 and 13) by Analysis of Circulating Fetal DNA in a Population of Pregnant Patients With Autoimmune Diseases"
Brief Title: "Circulating Fetal DNA, Pregnancy And Immune Diseases"
Acronym: AFFEPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CERBA laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180669; 2019-A01827-50 (Other: IDRCB number)
Record Dates: First submitted 2019-09-17; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-09

CONDITIONS: Autoimmune Diseases; Pregnancy
Keywords: autoimmune disease; pregnancy; free fetal DNA circulant
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed group (patient with an autoimmunise disease) (Experimental): Any patient with an autoimmune disease followed at one of the 14 centres who wants to be screened for T21.
  Interventions: Biological: the detection of the risk of fetal trisomy 21 by blood tests : free fetal DNA circulant analysis
- Non Exposed group (patient without an autoimmunise disease) (Other)
  Interventions: Biological: the detection of the risk of fetal trisomy 21 by blood tests : free fetal DNA circulant analysis

INTERVENTIONS:
Biological: the detection of the risk of fetal trisomy 21 by blood tests : free fetal DNA circulant analysis — The detection of the risk of fetal trisomy 21 by blood tests by 2 tests : free fetal DNA circulant analysis and first trimester serum screening

SUMMARY:
In the plasma of any pregnant patient circulates DNA (also called circulating free DNA). The vast majority of this circulating free DNA is of maternal origin and about 10% is of fetal origin (fetal circulating free DNA). This percentage of fetal circulating free DNA (corresponding to the fetal fraction) increases with gestation.

The pathophysiological hypothesis of this research is that there is a change in the fetal fraction (FF) of fetal circulating free DNA in patients with autoimmune disease (AID). The underlying mechanism would be a massive release of maternal cfDNA responsible for a dilution of fetal cfDNA. This dilution of fetal cfDNA would result in a decrease in the estimate of the foetal fraction of circulating free DNA. However, when the foetal fraction of circulating free DNA is insufficient (4% most often), screening for Trisomy 21 (T21) by fetal circulating free DNA becomes uninterpretable (NC for "non-contributory" result), and cannot be used to assess the risk of T21. In this case, the dose of fetal circulating free DNA can be performed again after 15 days, as the amount of fetal circulating free DNA increases with gestation. In a small number of cases the result will remain NC.

As tests using DNA are becoming more widespread, it is important to prospectively evaluate the results of these tests in the population of patients with AID, which represents about 3 to 5% of pregnant women.

DETAILED DESCRIPTION:
Circulating fetal DNA (cfDNA) in maternal blood is now routinely used for prenatal screening for Down syndrome 21 (T21). In about 1% of cases, the test result is not contributory (NC). The investigator's team recently found, in a retrospective study, an association between the existence of an autoimmune disease (AID) and a high risk of NC. However, this was only a subgroup analysis, requiring confirmation by a dedicated study. Tests using deoxyribonucleic Care (dNCare) are becoming more widespread, so it is important to prospectively evaluate the results of these tests in the population of patients with AID, which represents about 3 to 5% of pregnant women.

The main objective of this study is to compare the rate of NC in a population of patients with DIA to that of a population of patients without MAI when screened for T21 by the cfDNA study in the first trimester of pregnancy.

The secondary objectives are :

* To assess the performance of fetal cfDNA for T21 screening in the population of PATIENTS with AID and to compare them with performance in the non-auto immune disease population.
* To assess the performance of the combined first trimester screening for T21 screening and compare it with those of fetal cfDNA in the population of patients with AID.
* In patients with an NC result, analysis of the distribution of fetal fractions according to the presence and severity of maternal autoimmune pathologies. The distribution will be compared to that of the control population.
* To assess the association between fetal fraction and the occurrence of vascular complications of pregnancy in both groups with and without auto immune disease.

AFFEPI is a prospective multicenter, interventional, exposed/non-exposed cohort study

There are two group :

Exposed group: Any patient with a auto immune disease followed at one of the 14 centres who wants to be screened for T21.

Unexposed group: Patients who do not carry an auto immune disease identified at the interview (no history of auto immune disease; no symptoms suggestive of a auto immune disease).

ELIGIBILITY:
Inclusion Criteria:

Patients in the exposed group:

* Single-fetal pregnancy with a term between 11 and 13-6 weeks of amenorrhea (SA) from spontaneous pregnancy or by medical assistance to procreation.
* Age ≥ 18 years
* Affiliated with a social security or beneficiary scheme
* Desire for natal screening of T21, not yet realized
* Patient with a condition on the following list: [see Chapter 7.2]

Patients in the unexposed group:

* Single-fetal pregnancy with a term between 11 and 13-6 weeks of amenorrhea (SA) from spontaneous pregnancy or by medical assistance to procreation.
* Age ≥ 18 years
* Affiliated with a social security or beneficiary scheme
* Desire for natal screening of T21, not yet realized
* No pathology that meets the list mentioned in the above section
* Clinically asymptomatic patient with no clinical symptoms suggestive of AID: arthralgias, skin or mucous disease, dry syndrome, Raynaud syndrome, purpura.
* Patient respecting frequency pairing

Exclusion Criteria:

* BMI > 35 kg/cm2
* Multiple pregnancy
* No first trimester ultrasound (between 11 and 13-6 SA)
* Screening for unwanted T21
* Patients already included in an interventional research protocol
* Morphological abnormalities on first trimester ultrasound and/or nucal clarity - 3.5mm
* Patient under the protection of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant population
Enrollment: 320 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The number of inconclusive results of the free circulating fetal DNA test | maximum 15 days after inclusion if the result of the initial analysis is inconclusive. Or maximum 30 days after inclusion if the analysis is realized a second time
  The detection of the risk of fetal trisomy 21 by 2 blood tests : free circulating analysis fetal DNA and first trimester serum screening. A result of the free fetal DNA circulant test is rendered as inconclusive when the fetal fraction is strictly less than 4% or the result of the z-scores is not interpretable

SECONDARY OUTCOMES:
Performance (ability to detect the risk) of fetal DNA for T21 screening in the auto immune disease population. and To compare them with the non-auto immune disease population. | maximum 15 days after inclusion if the result of the initial analysis is inconclusive, or maximum 30 days after inclusion if the analysis is realized a second time
  The results of free circulating fetal DNA analysis and first trimester serum screening for T21 screening
Performance (ability to detect the risk) of the combined first trimester serum screening for T21 screening and compare it with those of fetal DNA in auto immune disease population. | maximum 15 days after inclusion if the result of the initial analysis is inconclusive, or maximum 30 days after inclusion if the analysis is realized a second time
  The results of free circulating fetal DNA analysis and first trimester serum screening for T21 screening
Distribution of fetal fractions according to the presence and severity of maternal autoimmune pathology | maximum 15 days after inclusion if the result of the initial analysis is inconclusive, or maximum 30 days after inclusion if the analysis is realized a second time
  Distribution of the results of free circulating fetal DNA analysis and first trimester serum screening for T21 screening in the group of patient with autoimmune disease
Association between fetal fraction and the occurrence of vascular complications of pregnancy in both groups with and without auto immune disease. | maximum 15 days after inclusion if the result of the initial analysis is inconclusive, or after inclusion if the analysis is realized a second time
  The detection of the risk of fetal trisomy 21 : Free circulating fetal DNA analysis and first trimester serum screening

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Antoine Béclère, Clamart, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No